CLINICAL TRIAL: NCT03025880
Title: A Multicenter Phase II Trial to Evaluate the Efficacy and Safety of Pembrolizumab and Gemcitabine in Patients With HER2-negative Advanced Breast Cancer (ABC) "PANGEA-Breast"
Brief Title: Trial to Evaluate Efficacy and Safety of Pembrolizumab and Gemcitabine in HER2-negative ABC
Acronym: PANGEA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Spanish Breast Cancer Research Group (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GEICAM/2015-04; 2016-001779-54 (EudraCT Number)
Record Dates: First submitted 2017-01-11; First posted 2017-01-20 (Estimated); Results first posted 2023-01-10 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Advanced Breast Cancer
Keywords: Advanced Breast Cancer; Pembrolizumab; HER2-negative
MeSH Terms: interventions — pembrolizumab; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single arm (Experimental): Eligible patients will be enrolled and treated with Pembrolizumab (P) at a dose of 200mg as an intravenous (IV) infusion on day 1 of each 21-day cycle in combination with Gemcitabine (G) at a dose of 1,250mg/m2 or 1,000mg/m2 (this dose will be explored in combination with P in the initial exploratory run-in-phase if necessary) as a IV infusion on day 1 and 8 of each 21-day cycle.
  Treatment will be repeated on day 1 of each 21-day cycle until objective disease progression, clinical progression (under investigator criteria), unacceptable toxicity, death or withdrawal of consent, whichever occurs first. An initial exploratory run-in-phase will be performed to test the safety of the combination and determine the Recommended Phase II Dose (RP2D) of G in combination with fixed doses of P.
  Interventions: Drug: Pembrolizumab; Drug: Gemcitabine

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab at a dose of 200mg as an intravenous (IV) 30 minutes infusion on day 1 of each 21-day cycle. Treatment will be repeated on day 1 of each 21-day cycle until objective disease progression, clinical progression (under investigator criteria), unacceptable toxicity, death or withdrawal of consent, whichever occurs first. Patients completing 24 months of uninterrupted treatment with pembrolizumab or 35 administrations of study medication will stop pembrolizumab treatment (though may continue with gemcitabine). Subjects who stop pembrolizumab after 24 months may be eligible for up to one year of additional pembrolizumab treatment if they progress after stopping it.
  Other Names: Keytruda
Drug: Gemcitabine — Gemcitabine at a dose of 1,250mg/m2 as an intravenous (IV) 60 minutes infusion on day 1 and 8 of each 21-day cycle. Treatment will be repeated on day 1 of each 21-day cycle until objective disease progression, clinical progression (under investigator criteria), unacceptable toxicity, death or withdrawal of consent, whichever occurs first.
  Other Names: Gemzar

SUMMARY:
Study Design and Treatment:

This is a multicenter phase II trial, with an initial exploratory run-in-phase, to evaluate the efficacy and safety of pembrolizumab in combination with gemcitabine in patients with HER2-negative ABC that have previously received anthracyclines and taxanes (unless clinically contraindicated). In hormone receptor positive patients, previous treatment with 2 or more lines of hormone therapy will also be required. Patients must have at least one measurable lesion that can be accurately assessed at baseline and is suitable for repeated assessment by CT, MRI or plan X-ray. Approximately 53 patients (up to a maximum of 65 patients depending on the results of the run-in-phase) will be included in this trial.

DETAILED DESCRIPTION:
Study Design and Treatment (continuation):

The study will include two cohorts of patients: i) Triple Negative and ii) Luminal A+B, with an approximate 1:1 distribution between both groups.

A safety dose testing or "run-in-phase", with a 6+6 design, in which toxicity will be evaluated within the first cycle, will be performed since pembrolizumab in combination with gemcitabine has not been previously tested. Initially 6 patients will be included in the study at dose level 0 (gemcitabine at a dose of 1,250mg/m2 as an IV infusion on day 1 and 8 of each 21-day cycle and pembrolizumab at a dose of 200mg as an IV infusion on day 1 of each 21-day cycle):

* If ≤ 2 patients experience Dose Limiting Toxicity (DLT), 6 additional patients will be included at the current dose level. If there is a confirmation of this dose to be safe (≤ 3 patients experiencing DLT), this will be considered the RP2D and it will be used for the following recruited patients.
* If ≥ 3 patients experience DLT within the first 6 patients, or ≥ 4 within the first 12 patients included at dose level 0, a de-escalation to dose level -1 (gemcitabine at a dose of 1,000mg/m2 as an IV infusion on day 1 and 8 of each 21-day cycle and pembrolizumab at a dose of 200mg as an IV infusion on day 1 of each 21-day cycle) will be performed. In this case, a group of 12 additional patients will be included at dose level -1, if ≥ 4 experience DLT, this combination will be considered too toxic and the study will be stopped. If ≤ 3 experience DLT with this combination, this will be considered the RP2D and it will be used for the following recruited patients.

Initially 3 patients will be allowed for inclusion simultaneously. These 3 patients will be followed closely during the first cycle to observe the occurrence of any DLT. At the times these 3 patients are completing the first cycle, the next 3 patients will be included one by one, until the first cohort is completed.

If none of these 6 patients have a DLT, up to 4 patients will be allowed for inclusion from the second cohort of 6 patients; they will follow the same procedure as in the first cohort. If one of these patients from the second cohort has a DLT, the inclusion will be in smaller groups (with a maximum number of 4 patients with DLT) and following the same procedure as in the first cohort of 6 patients.

An internal committee will periodically review the safety data in order to take the decision to maintain or decrease the dose level. This internal committee will consist of the chief investigator, the Spanish Breast Cancer Research Group Scientific Director and the study statistician. The meetings will be performed by teleconference to take these decisions as quickly as possible once the last patient finishes the first cycle of treatment. Other meetings will be considered ad-hoc whenever necessary (i.e when new DLTs appear).

Patients included in the run-in-phase at the same dose than that in the phase II will be considered for the phase II analysis.

Study Drug/Medication:

Eligible patients will be enrolled and treated with:

Pembrolizumab at a dose of 200mg as an intravenous (IV) infusion on day 1 of each 21-day cycle.

in combination with Gemcitabine at a dose of 1,250mg/m2 or 1,000mg/m2 (this dose will be explored in combination with pembrolizumab in the initial exploratory run-in-phase if necessary) as an intravenous (IV) infusion on day 1 and 8 of each 21-day cycle.

Treatment will be repeated on day 1 of each 21-day cycle until objective disease progression, clinical progression (under investigator criteria), unacceptable toxicity, death or withdrawal of consent, whichever occurs first. Patients completing 24 months of uninterrupted treatment with pembrolizumab or 35 administrations of study medication will stop pembrolizumab treatment (though may continue with gemcitabine). Subjects who stop pembrolizumab after 24 months may be eligible for up to one year of additional pembrolizumab treatment if they progress after stopping it.

An initial exploratory run-in-phase will be performed to test the safety of the combination and determine the Recommended Phase II Dose (RP2D) of gemcitabine in combination with fixed doses of pembrolizumab.

Primary Objective:

* Run-in-phase: To determine the Recommended Phase II Dose (RP2D) of gemcitabine in combination with fixed doses of pembrolizumab.
* Phase II: To assess the efficacy of pembrolizumab in combination with gemcitabine in terms of Objective Response Rate (ORR) in patients with HER2-negative ABC.

Primary End-point:

* Run-in-phase: To determine the incidence rate of Dose Limiting Toxicity (DLT) within the first cycle of the combination.
* Phase II: Objective Response Rate (ORR) is defined as Complete Response (CR) plus Partial Response (PR) according to Response Evaluation Criteria in Solid Tumours (RECIST) version 1.1.

Secondary Objectives:

The following secondary objectives will be studied:

* To assess other efficacy measures of the combination in patients included in the phase II (including those in the run-in-phase at the same dose that in the phase II).
* To determine safety and tolerability of the combination in all patients included in the study.

Secondary End-points:

The following secondary end-points will be studied:

* Efficacy:

  * Progression-Free Survival (PFS) assessed according to RECIST version 1.1 by the investigator.
  * Clinical Benefit Rate (CBR) defined as Complete Response (CR) plus Partial Response (PR) plus Stable Disease (SD) lasting ≥ 24 weeks according to RECIST version 1.1.
  * Response Duration (RD) assessed according to RECIST version 1.1.
  * Overall Survival (OS). With special interest on long term responders (i.e. alive and without disease progression after 24 months of study treatment).
* Safety will be assessed by standard clinical and laboratory tests (haematology, serum chemistry). Adverse Events (AE) grade will be defined by the NCI CTCAE (National Cancer Institute Common Terminology Criteria for Adverse Events) version 4.0.

Exploratory Objectives:

The following exploratory objectives will be studied in all patients included in the study unless otherwise specified:

* To assess other efficacy measures of the combination based on immune-related (ir) response criteria in patients included in the phase II (including those in the run-in-phase at the same dose that in the phase II).
* To search for tumour tissue and peripheral blood biomarkers of clinical activity.
* To compare biomarkers data from cohorts of healthy volunteers (if available) with data from patients included in the study.

Exploratory End-points:

The following exploratory end-points will be studied:

* Efficacy:

  * ORR is defined as immune-related Complete Response (irCR) plus immune-related Partial Response (irPR) according to immune-related RECIST (irRECIST).
  * Progression-Free Survival (PFS) assessed according to irRECIST by the investigator.
  * Clinical Benefit Rate (CBR) defined as irCR plus irPR plus immune-related Stable Disease (irSD) lasting ≥ 24 weeks according to irRECIST.
  * Response Duration (RD) assessed according to irRECIST.
* A set of immune biomarkers will be analysed and correlated with evolution of the disease and efficacy of pembrolizumab in combination with gemcitabine (ORR and other efficacy end-points: PFS, CBR and RD), paying special attention to long term responders.
* This set of immune biomarkers will be compared with those from healthy volunteers (if available).

Study population:

Patients with HER2-negative advanced breast cancer.

Justification of Sample size determination:

A Simon's minimax two-stage design will be employed with the possibility of stopping early due to lack of response. Results from previous studies showed that gemcitabine produced a response rate of around 20%, this will be our expected H0. With the combination of pembrolizumab and gemcitabine, we expect to increase this rate to 35% what will be our H1 (an absolute increase of 15%), with an alpha error of 0.05 and a statistical power of 80%, we will need to include 53 evaluable patients in this trial. The first stage will include 31 evaluable patients, if at least 7 present a response, recruitment will continue to include the 53 evaluable patients. The null hypothesis of H0=20% will be rejected if 16 or more responses are observed in 53 patients.

Statistical Analyses:

Demographics and Baseline Characteristics: Standard descriptive statistics, such as the mean, median, range and proportion, will be used to summarize the patient sample and to estimate parameters of interest.

Safety Analyses: AEs and Serious Adverse Events (SAE) will be reported in frequency tables (overall and by intensity). The safety analysis will be performed in the population that has received at least one dose of any of the study drugs/medications.

Efficacy Analyses: All efficacy endpoints will be evaluated in the Per-protocol and Intent to treat (ITT) populations.

Biomarker analysis:The biomarker analysis will be exploratory and descriptive. For continuous variables, mean, standard deviation, median, minimum and maximum values will be provided. Categorical variables will be summarized by numbers and proportions. Biomarker endpoints will be evaluated in all patients enrolled in the study with available samples.

Study Duration:

The end date of study is date of last patient´s death or the date when there is sufficient data to achieve the primary and secondary objectives and all patients have ended the study treatment, whichever comes first.

Performing exploratory objectives will be independent of the date of the end of the study.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has signed and dated the informed consent document and it has been obtained before conducting any procedure specifically for the study.
2. Female ≥ 18 years of age on day of signing informed consent.
3. Histological/cytological confirmation of breast cancer with evidence of advanced disease, not amenable to resection or radiation therapy with curative intent.
4. Documented luminal A, luminal B (HER2-negative) or triple negative disease by immunohistochemistry (IHQ) and/or in situ hybridization (FISH/CISH/SISH) based on local testing on the most recent tumour biopsy defined as follows:

   Luminal A: tumour with positive oestrogen receptor (ER) status (≥1% of tumour cells with ER expression) and HER2-negative status (IHQ score 0/1+ or negative by in situ hybridization defined as a HER2/chromosome enumeration probe 17 (CEP17) ratio < 2 or for single probe assessment a HER2 copy number < 4) and high progesterone receptor (PgR) (≥ 20% of tumour cells with PgR expression) and low Ki67 (< 14%).

   Luminal B (HER2-negative): tumour with positive ER status (≥1% of tumour cells with ER expression) and HER2-negative status (IHQ score 0/1+ or negative by in situ hybridization defined as a HER2/CEP17 ratio < 2 or for single probe assessment a HER2 copy number < 4) and either low or negative PgR (< 20% of tumour cells with PgR expression) and/or high Ki67 (≥ 14%).

   Triple negative: tumour with negative hormone receptor status (<1% of tumour cells with ER and PgR expression) and HER2-negative status (IHQ score 0/1+ or negative by in situ hybridization defined as a HER2/CEP17 ratio < 2 or for single probe assessment a HER2 copy number < 4).
5. Have at least one unidimensionally measurable lesion by RECIST 1.1.
6. Patient agrees to the collection of a metastatic tumor sample (biopsy) at the time of inclusion and at progression (whenever possible).
7. Have a performance status of 0, 1 or 2 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
8. Demonstrate adequate organ function as follows (all screening labs should be performed within 7 days of study treatment initiation):

   Bone marrow:

   Absolute Neutrophil Count (ANC) ≥ 1,500/mm3 (1.5x109/l) Platelets ≥ 100,000/mm3 (100x109/l) Hemoglobin ≥ 9g/dl or ≥ 5.6 mmol/l without transfusion or erythropoietin (EPO) dependency (within 7 days of assessment)

   Hepatic:

   Serum total bilirubin ≤ 1.5 x Upper Limit of Normal (ULN) Alkaline Phosphatase ≤ 2.5 x ULN Aspartate aminotransferase (AST) (SGOT) and Alanine aminotransferase (ALT) (SGPT) ≤ 2.5 x ULN or ≤ 5 x ULN for patients with liver metastases Albumin ≥ 2.5 g/dl

   Renal:

   Serum creatinine ≤ 1.5 x ULN or creatinine clearance ≥ 60 ml/min for patients with creatinine levels > 1.5 x ULN

   Coagulation:

   International Normalized Ratio (INR) or Prothrombin Time (PT) ≤ 1.5 x ULN unless patient is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants.

   Activated Partial Thromboplastin Time (aPTT) ≤ 1.5 x ULN unless patient is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants.
9. Prior treatment with anthracyclines and taxanes (unless clinically contraindicated) and two or more prior lines of hormone therapy in hormone receptor positive disease.
10. At least 3 months life expectancy.
11. Patient of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study drug/medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
12. Patients of childbearing potential (see section 4.4. for definition) must be willing to use an adequate method of contraception as outlined in Section 4.4. - Contraception, for the course of the study through 120 days after the last dose of study medication.

    Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
13. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests and other study procedures.

Exclusion Criteria:

1. HER2-positive disease by immunohistochemistry or in situ hybridation (FISH-SISH-CISH).
2. Patient is currently participating or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of study drug/medication.
3. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study day 1 or who has not recovered (i.e., ≤ grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
4. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study day 1 or who has not recovered (i.e., ≤ grade 1 or at baseline) from adverse events due to a previously administered agent.

   * Note: Patients with ≤ grade 2 neuropathy are an exception to this criterion and may qualify for the study.
   * Note: If patient received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
5. Has received prior therapy with an anti-Programmed death-1 (PD), anti-PD-L1, or anti-PD-L2 agent.
6. Has received a live vaccine within 30 days of planned start of study therapy.

   o Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however, intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed.
7. Has hypersensitivity to pembrolizumab, gemcitabine or any of theirs excipients.
8. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and all neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
9. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug/medication.
10. Has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
11. Has a current or prior malignancy within the previous 5 years (other than breast cancer or adequately treated basal cell or squamous cell carcinoma of the skin or in-situ carcinoma of the cervix).
12. Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
13. Has an active infection requiring systemic therapy.
14. Has a known history of active Tuberculosis Bacillus (TB) or Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies) or a known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., hepatitis C virus (HCV) RNA [qualitative] is detected).
15. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating investigator.
16. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
17. Patient is pregnant or breastfeeding, or expecting to conceive within the projected duration of the trial, starting with the baseline visit through 120 days after the last dose of trial treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-06-28 (Actual); Primary Completion 2019-06-03 (Actual); Study Completion 2021-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Hospital Universitario Virgen Macarena
Locations (9):
- Spain (9):
  - Institut Català d'Oncologia. Hospital Universitario Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Canary Islands
  - Hospital Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Clínica Universitaria de Navarra, Pamplona, Navarre
  - Centro Oncológico de Galicia, A Coruña
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Clínico Universitario San Carlos, Madrid
  - Hospital Universitario Virgen de la Macarena, Seville
  - Hospital Clínico Universitario de Zaragoza "Lozano Blesa", Zaragoza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] de la Cruz-Merino L, Gion M, Cruz J, Alonso-Romero JL, Quiroga V, Moreno F, Andres R, Santisteban M, Ramos M, Holgado E, Cortes J, Lopez-Miranda E, Cortes A, Henao F, Palazon-Carrion N, Rodriguez LM, Ceballos I, Soto A, Puertes A, Casas M, Benito S, Chiesa M, Bezares S, Caballero R, Jimenez-Cortegana C, Sanchez-Margalet V, Rojo F. Pembrolizumab in combination with gemcitabine for patients with HER2-negative advanced breast cancer: GEICAM/2015-04 (PANGEA-Breast) study. BMC Cancer. 2022 Dec 3;22(1):1258. doi: 10.1186/s12885-022-10363-3. PMID 36463104
- [Result] de la Cruz-Merino L, Gion M, Cruz-Jurado J, Quiroga V, Andres R, Moreno F, Alonso-Romero JL, Ramos M, Holgado E, Cortes J, Lopez-Miranda E, Henao-Carrasco F, Palazon-Carrion N, Rodriguez LM, Ceballos I, Casas M, Benito S, Chiesa M, Bezares S, Caballero R, Jimenez-Cortegana C, Sanchez-Margalet V, Rojo F. Pembrolizumab Plus Gemcitabine in the Subset of Triple-Negative Advanced Breast Cancer Patients in the GEICAM/2015-04 (PANGEA-Breast) Study. Cancers (Basel). 2021 Oct 29;13(21):5432. doi: 10.3390/cancers13215432. PMID 34771596
- See also: GEICAM is a Spanish Breast Cancer Research Group — http://www.geicam.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Fourteen patients were enrolled at the Run-in phase, receiving at least one cycle of the combination. All patients were included at Dose Level (DL) 0. Twenty-two patients were included at the phase II.
Groups:
- Run-in Phase Dose Level 0: Eligible patients were enrolled and treated with Pembrolizumab (P) at a dose of 200mg as an intravenous (IV) infusion on day 1 of each 21-day cycle in combination with Gemcitabine (G) at a dose of 1,250mg/m2 (Dose Level 0) or 1,000mg/m2 (Dose Level -1) as a IV infusion on day 1 and 8 of each 21-day cycle.
  Treatment will be repeated on day 1 of each 21-day cycle until objective disease progression, clinical progression (under investigator criteria), unacceptable toxicity, death or withdrawal of consent, whichever occurs first.
  An initial exploratory run-in-phase will be performed to test the safety of the combination and determine the Recommended Phase II Dose (RP2D) of G in combination with fixed doses of P.
- Phase II: Eligible patients were enrolled and treated with Pembrolizumab (P) at a dose of 200mg as an intravenous (IV) infusion on day 1 of each 21-day cycle in combination with Gemcitabine (G) at a dose of 1,250mg/m2 (Recommended Phase II Dose (RP2D) from the run-in phase) as a IV infusion on day 1 and 8 of each 21-day cycle.
  Treatment will be repeated on day 1 of each 21-day cycle until objective disease progression, clinical progression (under investigator criteria), unacceptable toxicity, death or withdrawal of consent, whichever occurs first.
Period: Overall Study
Arm/Group | Run-in Phase Dose Level 0 | Phase II
Started | 14 | 22
Completed | 0 | 0
Not Completed | 14 | 22
Not completed — Adverse Event | 1 | 0
Not completed — Death | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Progressive Disease | 12 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Run-in Phase Dose Level 0 | Phase II | Total
Number analyzed (Participants) | 14 | 22 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 19 | 33
  >=65 years | 0 | 3 | 3
Age, Continuous [Median (Standard Deviation); unit: years] | 48.5 (8) | 56 (12.19) | 51.5 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 22 | 36
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 14 | 22 | 36
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Spain | 14 | 22 | 36
Menopause Status [Count of Participants; unit: Participants]
  Postmenopausal | 10 | 16 | 26
  Premenopausal | 4 | 6 | 10
Eastern Cooperative Oncology Group (ECOG) status [Count of Participants; unit: Participants] — ECOG score runs from 0 to 5, with 0 denoting perfect health and 5 death. 0 - Asymptomatic
  1. - Symptomatic but completely ambulatory
  2. - Symptomatic, <50% in bed during the day
  3. - Symptomatic, >50% in bed, but not bedbound
  4. - Bedbound
  5. - Death
  Participants
    ECOG 0 | 7 | 16 | 23
    ECOG 1 | 6 | 6 | 12
    ECOG 2 | 1 | 0 | 1
Type of Disease for Cohort Purposes [Count of Participants; unit: Participants] — Luminal A: estrogen-receptor (ER) and/or progesterone-receptor (PR) positive, Human Epidermal Growth Factor Receptor 2 (HER2) negative, low levels of Ki67. Luminal A are low-grade, tend to grow slowly and have the best prognosis.
  Luminal B: ER and/or PR positive, and HER2 positive or HER2 negative with high levels of Ki67. Luminal B grow faster than luminal A and their prognosis is worse.
  Triple-negative (TN): negative for ER, PR, and HER2. Is more aggressive and have poorer prognosis than Luminal due to there are fewer targeted medicines that treat TN.
  Participants
    Triple negative | 9 | 12 | 21
    Luminal A+B | 5 | 10 | 15
Ki67 cut-off 20% [Count of Participants; unit: Participants] — Ki67 is a protein found in the nucleus of cells when they divide. Ki67 determines the proliferation rate. Tumors with high proliferation rates (> 20%) have a worse prognosis.
  Participants
    Ki67 <20% | 1 | 4 | 5
    Ki67 >=20% | 8 | 13 | 21
    Ki67 Not Available/Not Done | 5 | 5 | 10
Histopathologic Type [Count of Participants; unit: Participants]
  Ductal | 13 | 20 | 33
  Lobular | 1 | 1 | 2
  Other: Squamous Invasive Cancer | 0 | 1 | 1
Histologic Grade [Count of Participants; unit: Participants] — Cancer cells are given a Grade (G) when they are removed from the breast and checked under a microscope. The G is based on how much the cancer cells look like normal cells.
  G1 or well differentiated (score 3, 4, or 5): cells are slower-growing, and look more like normal breast tissue.
  G2 or moderately differentiated (score 6, 7): cells are growing at a speed of and look like cells somewhere between G1 and 3.
  G3 or poorly differentiated (score 8, 9): cells look very different from normal and will probably grow and spread faster.
  Participants
    Grade 1 | 0 | 1 | 1
    Grade 2 | 4 | 10 | 14
    Grade 3 | 6 | 10 | 16
    Unknown | 1 | 0 | 1
    Not done | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicity (DLT) Within the First Cycle
Description: DLT was defined as the occurrence of any of the following adverse events (AE) or abnormal laboratory value (graded according to the NCI Common Terminology Criteria for AE (CTCAE) version 4.0), assessed as possibly, probably or definitively related to study drug/medication, occurring within the first cycle of study treatment: any Grade 4 thrombocytopenia or neutropenia lasting > 7 days; episcleritis, uveitis, or iritis of Grade 2 or higher, any Grade 4 toxicity, any Grade 3 toxicity EXCLUDING: nausea, vomiting, or diarrhea controlled by medical intervention within 72 hours, grade 3 rash in the absence of desquamation, no mucosal involvement, does not require steroids, and resolves to Grade 1 by the next scheduled dose of pembrolizumab, transient Grade 3 Aspartate Transaminase (AST) or Alanine Transaminase (ALT) elevation, defined as no more than 3 days with or without steroid use, discontinuation or delay of more than 2 weeks of any study drug/medication due to treatment-related AE.
Time Frame: Up to cycle 1
Population: There was no need to explore the Dose Level -1 (Pembrolizumab 200mg intravenous (IV) infusion on day 1 of each 21-day cycle in combination with Gemcitabine 1,000mg/m2 as a IV infusion on day 1 and 8 of each 21-day cycle.
Measure: Count of Participants; unit: Participants
Groups:
- Run-in Phase Dose Level 0: Eligible patients were enrolled and treated with Pembrolizumab (P) at a dose of 200mg as an intravenous (IV) infusion on day 1 of each 21-day cycle in combination with Gemcitabine (G) at a dose of 1,250mg/m2 (Dose Level 0) as a IV infusion on day 1 and 8 of each 21-day cycle.
  Treatment will be repeated on day 1 of each 21-day cycle until objective disease progression, clinical progression (under investigator criteria), unacceptable toxicity, death or withdrawal of consent, whichever occurs first.
Arm/Group | Run-in Phase Dose Level 0
Number analyzed (Participants) | 14
Participants | 1

2. Primary Outcome: Recommended Phase II Dose (RP2D) of Gemcitabine in Combination With Pembrolizumab
Description: The RP2D was decided by the internal committee taken into consideration the information obtained in the study and based on the number of DLT.
Time Frame: Up to cycle 1
Population: Run in phase population
Measure: Number; unit: mg/m2
Arm/Group | Run-in Phase Dose Level 0
Number analyzed (Participants) | 14
mg/m2 | 1250

3. Primary Outcome: Objective Response Rate (ORR)
Description: Tumor response was assessed using Response Evaluation Criteria In Solid Tumors Criteria (RECIST 1.1). ORR is defined as the percentage of patients with a Complete Response (CR) or Partial Response (PR) out of the patients from the efficacy population. Per RECIST, CR is defined as the disappearance of all target lesions; PR is defined as an >=30% decrease in the sum of the longest diameter of target lesions.
Time Frame: Through study treatment, and average of 3 months
Population: Efficacy population: patients that had measurable disease, had received at least one dose of study treatment and had at least one tumor response assessment (unless progression or death or unacceptable toxicity before the first tumor response assessment) and without certain major protocol deviations according to the protocol deviation manual.
Measure: Count of Participants; unit: Participants
Groups:
- Run-in Phase Plus Phase II: Patients included in the run-in-phase at the same dose that in the phase II (DL0) were included on the analysis.
Arm/Group | Run-in Phase Dose Level 0 | Phase II | Run-in Phase Plus Phase II
Number analyzed (Participants) | 13 | 20 | 33
Participants | 0 | 5 | 5

4. Secondary Outcome: Progression-Free Survival (PFS)
Description: Tumor response was assessed using Response Evaluation Criteria In Solid Tumors Criteria (RECIST 1.1). PFS is defined as the time from enrollment to the first documented progression disease (PD), or death from any cause, whichever occurs first. PD is defined using RECIST, as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: Through study treatment, and average of 3 months
Population: Efficacy population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Run-in Phase Dose Level 0 | Phase II | Run-in Phase Plus Phase II
Number analyzed (Participants) | 13 | 20 | 33
Months | 3.1 [0.9 to 5.4] | 2.6 [1.9 to 6.1] | 3.1 [2 to 4.3]

5. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: Tumor response was assessed using Response Evaluation Criteria In Solid Tumors Criteria (RECIST 1.1) criteria. CBR was defined as the percentage of patients with a Complete Response (CR) or Partial Response (PR) plus stable disease (SD) out of the efficacy population. Per RECIST, CR is defined as the disappearance of all target lesions; PR is defined as an >=30% decrease in the sum of the longest diameter of target lesions; SD is defined as a failure to meet criteria for CR or PR in the absence of progressive disease. Overall Response (OR) = CR + PR.
Time Frame: Through study treatment, and average of 3 months
Population: Efficacy population
Measure: Count of Participants; unit: Participants
Arm/Group | Run-in Phase Dose Level 0 | Phase II | Run-in Phase Plus Phase II
Number analyzed (Participants) | 13 | 20 | 33
Participants | 7 | 10 | 17

6. Secondary Outcome: Clinical Benefit Rate (CBR) at Least 24 Weeks
Description: Tumor response was assessed using Response Evaluation Criteria In Solid Tumors Criteria (RECIST 1.1) criteria. CBR was defined as the percentage of patients with a Complete Response (CR) or Partial Response (PR) plus stable disease (SD) lasting at least 24 months out of the efficacy population. Per RECIST, CR is defined as the disappearance of all target lesions; PR is defined as an >=30% decrease in the sum of the longest diameter of target lesions; SD is defined as a failure to meet criteria for CR or PR in the absence of progressive disease lasting at least 24 months. Overall Response (OR) = CR + PR.
Time Frame: 24 weeks
Population: Efficacy population
Measure: Count of Participants; unit: Participants
Arm/Group | Run-in Phase Dose Level 0 | Phase II | Run-in Phase Plus Phase II
Number analyzed (Participants) | 13 | 20 | 33
Participants | 1 | 5 | 6

7. Secondary Outcome: Response Duration (RD)
Description: Tumor response was assessed using Response Evaluation Criteria In Solid Tumors Criteria (RECIST 1.1) criteria. RD was defined as the time from the first documentation of objective tumor response (complete response (CR) or partial response (PR)) to the first documented progressive disease (PD), or to death due to any cause, whichever occurs first. Per RECIST, CR is defined as the disappearance of all target lesions; PR is defined as an >=30% decrease in the sum of the longest diameter of target lesions; PD is defined as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: Through study treatment, and average of 3 months
Population: There were only 5 Partial Responses on the phase II population.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Run-in Phase Dose Level 0 | Phase II | Run-in Phase Plus Phase II
Number analyzed (Participants) | 0 | 5 | 5
Months |  | 4.3 [2.3 to 7.4] | 4.3 [2.3 to 7.4]

8. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from the date of enrollment to the date of death from any cause.
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Run-in Phase Dose Level 0 | Phase II | Run-in Phase Plus Phase II
Number analyzed (Participants) | 13 | 20 | 33
Months | 6.1 [1.3 to 11.7] | 10.1 [7.3 to 17.7] | 8.7 [6.5 to 11.7]

9. Secondary Outcome: The Number of Participants Who Experienced Adverse Events (AE) Related to Study Treatment
Description: Safety assessments were performed at baseline and during the study: Vital signs assessments (blood pressure, pulse and body temperature), Laboratory assessments (hemoglobin, platelet count, White Blood Cell (WBC), Absolute Neutrophil Count (ANC) and Absolute Lymphocyte Count (ALC), albumin, alkaline phosphatase, alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin, serum creatinine, creatinine clearance (for patients with creatinine levels > 1.5 x ULN), glucose and urea, International Normalized Ratio (INR)/ Prothrombin time (PT) and activated partial thromboplastin time (aPTT), total or free triiodothyronine (T3 or FT3), free thyroxine (FT4) and Thyroid-stimulating hormone (TSH)) and Urinalysis. A baseline standard 12-lead electrocardiogram (ECG) was mandatory. AEs were graded according to NCI-CTCAE (National Cancer Institute Common Terminology Criteria for Adverse Events) version 4.03.
Time Frame: Through study treatment, and average of 3 months
Population: Safety population: patients who were enrolled and had have received at least one dose of the study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Run-in Phase Dose Level 0 | Phase II
Number analyzed (Participants) | 14 | 22
Participants | 8 | 17

10. Secondary Outcome: Immune-related Objective Response Rate (irORR)
Description: Tumor response was assessed using Immune-Related Response Evaluation Criteria In Solid Tumors Criteria (irRECIST v 1.0). irORR is defined as the percentage of patients with a Immune-Related Complete Response (irCR) or Immune-Related Partial Response (irPR) out of the patients from the efficacy population. Per irRECIST, irCR is defined as the disappearance of all measurable and non-measurable lesions, and lymph nodes must decrease to < 10 mm in short axis; irPR is defined as an >=30% decrease in total measured tumor burden relative to baseline; Immune-Related Overall Response (irOR) = irCR + irPR.
Time Frame: Through study treatment, and average of 3 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Run-in Phase Dose Level 0 | Phase II | Run-in Phase Plus Phase II
Number analyzed (Participants) | 13 | 20 | 33
Participants | 0 | 5 | 5

11. Secondary Outcome: Immune-related Progression-Free Survival (irPFS)
Description: Tumor response was assessed using Immune-Related Response Evaluation Criteria In Solid Tumors Criteria (irRECIST v 1.0). irPFS was defined as the time from enrollment to the first documented progressive disease (PD), or death from any cause, whichever occurs first. PD is defined by irRECIST, as a 20% increase and minimum 5 mm absolute increase in total measured tumor burden compared with nadir, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Through study treatment, and average of 3 months
Population: Efficacy population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Run-in Phase Dose Level 0 | Phase II | Run-in Phase Plus Phase II
Number analyzed (Participants) | 13 | 20 | 33
Months | 3.1 [1.3 to 7.7] | 2.6 [1.9 to 6.1] | 3.1 [2.0 to 5.4]

12. Secondary Outcome: Immune Related Clinical Benefit Rate (irCBR)
Description: Tumor response was assessed using Immune-Related Response Evaluation Criteria In Solid Tumors Criteria (irRECIST v 1.0). irCBR was defined as the percentage of patients with a Immune Related Complete Response (irCR) or Immune Related Partial Response (irPR) plus Immune Related Stable Disease (irSD) out of the efficacy population. Per irRECIST, irCR is defined as the disappearance of all measurable and non-measurable lesions, and lymph nodes must decrease to < 10 mm in short axis; irPR is defined as an >=30% decrease in total measured tumor burden relative to baseline; irSD is defined as a failure to meet criteria for irCR or irPR in the absence of progressive disease.
Time Frame: Through study treatment, and average of 3 months
Population: Efficacy population
Measure: Count of Participants; unit: Participants
Arm/Group | Run-in Phase Dose Level 0 | Phase II | Run-in Phase Plus Phase II
Number analyzed (Participants) | 13 | 20 | 33
Participants | 7 | 11 | 18

13. Secondary Outcome: Immune Related Clinical Benefit Rate (irCBR) at Least 24 Weeks
Description: Tumor response was assessed using Immune-Related Response Evaluation Criteria In Solid Tumors Criteria (irRECIST v 1.0). irCBR was defined as the percentage of patients with a Immune Related Complete Response (irCR) or Immune Related Partial Response (irPR) plus Immune Related stable disease (irSD) lasting at least 24 months out of the efficacy population. Per irRECIST, irCR is defined as the disappearance of all measurable and non-measurable lesions, and lymph nodes must decrease to < 10 mm in short axis; irPR is defined as an >=30% decrease in total measured tumor burden relative to baseline; irSD is defined as a failure to meet criteria for irCR or irPR in the absence of progressive disease at least 24 weeks.
Time Frame: Through study treatment, and average of 3 months
Population: Efficacy population
Measure: Count of Participants; unit: Participants
Arm/Group | Run-in Phase Dose Level 0 | Phase II | Run-in Phase Plus Phase II
Number analyzed (Participants) | 13 | 20 | 33
Participants | 1 | 5 | 6

14. Secondary Outcome: Immune Related Response Duration (irRD)
Description: Tumor response was assessed using Immune-Related Response Evaluation Criteria In Solid Tumors Criteria (irRECIST v 1.0). irRD was defined as the time from the first documentation of objective tumor response (immune related complete response (irCR) or immune related partial response (irPR)) to the first documented immune related progressive disease (irPD), or to death due to any cause, whichever occurs first. Per RECIST, irCR is defined as the disappearance of all measurable and non-measurable lesions, and lymph nodes must decrease to < 10 mm in short axis; irPR is defined as an >=30% decrease in total measured tumor burden relative to baseline; irPD is defined as a 20% increase and minimum 5 mm absolute increase in total measured tumor burden compared with nadir, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Through study treatment, and average of 3 months
Population: There were only 5 Partial Responses on the phase II population.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Run-in Phase Dose Level 0 | Phase II | Run-in Phase Plus Phase II
Number analyzed (Participants) | 0 | 5 | 5
Months |  | 4.3 [2.3 to 7.4] | 4.3 [2.3 to 7.4]

ADVERSE EVENTS:
Time Frame: AEs have been recorded through study treatment, an average of 3 months, and deaths have been recorded through study treatment and up to 2 years of follow up.
Description: AE were reported after Informed Consent Document (ICD) and before study drugs until approximately 30 days following the discontinuation of study treatment.
Arm/Group | Run-in Phase Dose Level 0 | Phase II
All-Cause Mortality (participants affected / at risk) | 12/14 | 19/22
Serious Adverse Events (participants affected / at risk) | 8/14 | 4/22
Other Adverse Events (participants affected / at risk) | 14/14 | 21/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Run-in Phase Dose Level 0 (N=14) | Phase II (N=22)
Abdominal sepsis (Infections and infestations) | 1 | 0
Bacterial pyelonephritis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Anemia Grade 2 and Platelet cound decreased Grade 2 (Investigations) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Neurological decompensation (Nervous system disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oedema peripheral (General disorders) | 0 | 1
Pancytopenia (Investigations) | 1 | 0
Intraabdominal bleeding (Investigations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Run-in Phase Dose Level 0 (N=14) | Phase II (N=22)
Neutrophil count decreased (Investigations) | 7 (53) | 15 (28)
Platelet count decreased (Investigations) | 8 (19) | 11 (18)
Alanine aminotransferase increased (Investigations) | 9 (24) | 11 (33)
Aspartate aminotransferase increased (Investigations) | 9 (30) | 13 (34)
Lymphocyte count decreased (Investigations) | 13 (101) | 12 (89)
White blood cell count decreased (Investigations) | 11 (82) | 18 (68)
Asthenia (General disorders) | 7 (9) | 14 (21)
Pyrexia (General disorders) | 4 (8) | 6 (7)
Anaemia (Blood and lymphatic system disorders) | 13 (136) | 21 (218)
Nausea (Gastrointestinal disorders) | 2 (4) | 6 (7)
Diarrhoea (Gastrointestinal disorders) | 2 (11) | 2 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (2) | 2 (3)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Alkaline phosphatase increased (Investigations) | 10 (46) | 14 (51)
INR increased (Investigations) | 2 (5) | 8 (33)
Blood bilirubin increased (Investigations) | 2 (4) | 2 (3)
Lymphocyte count increased (Investigations) | 1 (2) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 10 (30) | 9 (21)
Hyperglycemia (Metabolism and nutrition disorders) | 7 (15) | 4 (23)
Hypoglycemia (Metabolism and nutrition disorders) | 3 (6) | 2 (4)
Fatigue (General disorders) | 2 (2) | 0 (0)
Pain (General disorders) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (2) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (3)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Hypertension (Vascular disorders) | 0 (0) | 4 (7)
Hot flush (Vascular disorders) | 0 (0) | 2 (2)
Tachycardia (Cardiac disorders) | 2 (2) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (2)
Hypothyroidism (Endocrine disorders) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Albuminuria (Renal and urinary disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-03-19): https://cdn.clinicaltrials.gov/large-docs/80/NCT03025880/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-26): https://cdn.clinicaltrials.gov/large-docs/80/NCT03025880/SAP_001.pdf